CLINICAL TRIAL: NCT03293589
Title: Open Versus Endovascular Revascularization of Below-knee Arteries in Patients With End-stage Renal Disease and Critical Limb Ischemia
Brief Title: Open Versus Endovascular Revascularization in Patients With End-stage Renal Disease
Acronym: OERESRD
Status: Completed | Type: Observational
Sponsor: University Hospital Erlangen (Other)
Responsible Party: Principal Investigator, Alexander Meyer, MD, MD, University Hospital Erlangen
Other Study IDs: 00042158
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: End-stage Renal Disease; Critical Limb Ischemia
Keywords: end-stage renal disease; critical limb ischemia; surgical revascularisation; endovascular therapy
MeSH Terms: conditions — Kidney Failure, Chronic; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OR: patients treated with open revascularization
  Interventions: Procedure: open revascularization
- EVT: patients treated with endovascular revascularization
  Interventions: Procedure: endovascular revascularization

INTERVENTIONS:
Procedure: open revascularization — surgical revascularization (i.e. Bypass surgery)
  Groups: OR
Procedure: endovascular revascularization — endovascular revascularization (stent, ballon angioplasty)
  Groups: EVT

SUMMARY:
Treatment of patients with end-stage renal disease and critical limb ischemia still poses challenges to vascular medicine due to limited survival, comorbidities and infrapopliteal involvement of arteriosclerosis in these patients.

Most optimal vascular therapy mode has not been finally decided in these patients.

Therefore retrospective analysis of patients receiving open surgical and endovascular revascularisation was performed.

DETAILED DESCRIPTION:
Query of internal clinical database for identification of patients (2009-2017)with end-stage renal disease and critical limb ischemia, receiving either open surgical (Group I "OR") or endovascular revascularisation (Group II "EVT").

Furthermore, retrospective comparison as to morphological criteria (lesion length, peripheral run-off, plantar arch) and comorbidities.

Prospective follow-up of identified patients by means of telephone contacts and/or clinical examination of evaluation of Long-term outcome measures (Overall survival, Amputation-free survival, wound healing)

ELIGIBILITY:
Inclusion Criteria:

* presence of end-stage renal disease
* presence of critical limb ischemia (Ankle-brachial-index > 0.4 or presence of rest pain or ischemic ulcers or gangrene)
* revascularisation by means of Bypass or endovascular therapy

Exclusion Criteria:

* conservative Treatment
* non-atherosclerotic lesions
* coagulation disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: study Population comprises of all dialysis patients treated for critical limb ischemia by means of surgical or endiovascular Intervention at University Hospital Erlangen between 2009 and 2017
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Amputation free survival | 24 months
  Evaluation of limb salvage and survival as Composite endpoint

SECONDARY OUTCOMES:
Overall survival | 24 months
  Evaluation of Overall survival rate
Major Amputation | 24 months
  Evaluation of Major Amputation rate

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Meyer, MD, Principal Investigator — University Hospital Erlangen, Department of Vascular Sugery
Locations (1):
- University Hospital, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No